CLINICAL TRIAL: NCT03354052
Title: Efficacy of rTMS on Pain Following Stroke: a Pilot Randomized Control Trial.
Brief Title: Efficacy of rTMS on Pain Following Stroke.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Stroke_rTMS_Pain
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Stroke
Keywords: Pain; rTMS; Rehabilitation
MeSH Terms: conditions — Stroke; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-rTMS + Gloreha device (Experimental)
  Interventions: Device: Real-rTMS + Gloreha device
- Sham-rTMS + Gloreha device (Active Comparator)
  Interventions: Device: Sham-rTMS + Gloreha device

INTERVENTIONS:
Device: Real-rTMS + Gloreha device — The real rTMS will be delivered using a 8-shaped coil placed over the primary motor cortex (M1). The resting motor threshold (RMT) will be assessed at the place of the first dorsal interosseous (FDI) contralateral to the stimulated cortex. RMT of the FDI will be determined as the lowest strength of TMS needed to elicit 5 or more electromyographic responses ≥50 μV within 10 trials. Stimulation will be applied with frequency 10 Hz and intensity of 90% of RMT. Every session will last 15 minutes and includes 3000 pulses (30 trains of 10 seconds, following intertrain interval of 20 seconds). Rehabilitation programme will last 30 minutes and will be delivered using Gloreha® device, a proprioceptive stimulator under visual feedback. All the subjects enrolled will receive treatments for 2 weeks, 5 days per week.
  Arms: Real-rTMS + Gloreha device
Device: Sham-rTMS + Gloreha device — The sham rTMS will be delivered using a sham stimulator. All procedures will be performed as for the real treatment. Rehabilitation programme will last 30 minutes and will be delivered using Gloreha® device, a proprioceptive stimulator under visual feedback. All the subjects enrolled will receive treatments for 2 weeks, 5 days per week.
  Arms: Sham-rTMS + Gloreha device

SUMMARY:
Pain is a common symptom experienced by people following stroke and can significantly interfere with participation in the activities of daily living and adversely affect health-related quality of life. Repetitive Transcranial Magnetic Stimulation (rTMS) promotes the modulation of brain activity and its prolonged and continuous application can effect plastic modification. Combining rTMS with rehabilitation treatment for primary motor cortex activation (using Gloreha® device) may have effect in reducing pain in stroke survivors. This is a pilot randomized control trial to test the effects of rTMS in stroke-related pain rehabilitation, its efficacy on pain, upper limb function, sensory function and autonomy in daily livings activities. Furthermore, we will explore the effects on pressure pain threshold, cortical excitability and EEG recording.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of first stroke verified by brain imaging < 6 months
* pain defined as a constant or intermittent sensory symptom with unpleasant feelings or pain and a minimum score of 3 points on the Numeric Rating Scale (NRS) for pain perception

Exclusion Criteria:

* medical conditions likely to interfere with the ability to safely complete the study protocol
* cognitive functioning to give informed consent identified by a Mini-Mental Status Examination (MMSE) score ≥ 24/30
* intracranial metal implants
* history of seizures or epilepsy
* severe cardiopulmonary, renal, and hepatic diseases
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | Change measures (weeks: 0,2,6)
  Core outcome measure of pain intensity in pain treatments' clinical trials

SECONDARY OUTCOMES:
Neuropathic Pain Symptom Inventory (NPSI) | Change measures (weeks: 0,2,6)
  A self-questionnaire specifically designed to evaluate the different symptoms of neuropathic pain.
Short Form McGill Pain Questionnaire (SF-MPQ) | Change measures (weeks: 0,2,6)
  Assessment of sensory and affective dimensions of typical whole-body pain intensity.
Beck Depression Inventory II (BDI-II) | Change measures (weeks: 0,2,6)
  Assessment of severity of common depressive symptoms.
Erasmus MC modification to the (revised) Nottingham Sensory Assessment - Italian version (EmNSA-I) | Change measures (weeks: 0,2,6)
  Assessment of sensory function following brain injury.
Fugl-Meyer Assessment - Upper Extremity (FM-UE) | Change measures (weeks: 0,2,6)
  Assessment of upper limb function.
Barthel Index (BI) | Change measures (weeks: 0,2,6)
  Scale that measures disability or dependence in activities of daily living in stroke patients.
Pressure Pain Threshold (PPT) | Change measures (weeks: 0,2,6)
  PPT is measured to test presence of widespread pressure hyperalgesia as sign of abnormal pain processing.
Electroencephalography (EEG) recordings | Change measures (weeks: 0,2,6)
  EEG data will be recorded to test presence of particular brain activity in condition of pain.
Motor cortex excitability (single pulse TMS) | Change measures (weeks: 0,2,6)
  Single pulse TMS will be used to study cortical-spinal tract excitability in primary motor cortex (M1).

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Straudi, MD, PhD, Study Director — Ferrara Rehabilitation Hospital
Locations (1):
- Ferrara University Hospital, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No